CLINICAL TRIAL: NCT02412228
Title: BrUOG 299: Ixazomib, Oral Metronomic Cyclophosphamide and Dexamethasone for First-Line Treatment of Multiple Myeloma: A Phase II Brown University Oncology Group Study.
Brief Title: Ixazomib, Cyclophosphamide and Dexamethasone for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John L. Reagan (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Memorial Hospital of Rhode Island (Other)
Responsible Party: Sponsor-Investigator, John L. Reagan, Principal Investigator: Sponsor-Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 299
Record Dates: First submitted 2015-02-16; First posted 2015-04-09 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixazomib Regimen (Experimental): Cycle 1: Ixazomib: 4mg/day 1, 8, 15, Cyclophosphamide: 50 mg/day continuous daily, Dexamethasone: 20 mg/day 1, 8, 15 Cycles 2-6: Ixazomib: 4mg/day 1, 4, 8, 11, 15, 18, Cyclophosphamide: 50 mg/day continuous, daily, Dexamethasone: 20 mg/day 1, 4, 8, 11, 15, 18
  Maintenance:
  Ixazomib at 4 mg days 1, 8 and 15 of a 28 day cycle for 1 ½ years
  Interventions: Drug: Ixazomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Cycle 1:
  Ixazomib: 4mg/day 1, 8, 15
  Cycles 2-6:
  Ixazomib: 4mg/day 1, 4, 8, 11, 15, 18,
  Maintenance:
  Ixazomib at 4 mg days 1, 8 and 15 of a 28 day cycle for 1 ½ years
  Other Names: MLN978
Drug: Cyclophosphamide — Cycle 1:
  Cyclophosphamide: 50 mg/day continuous daily
  Cycles 2-6:
  Cyclophosphamide: 50 mg/day continuous daily
  Other Names: cytophosphane
Drug: Dexamethasone — Cycle 1:
  Dexamethasone: 20 mg/day 1, 8, 15
  Cycles 2-6:
  Dexamethasone: 20 mg/day 1, 4, 8, 11, 15, 18
  Other Names: Ozurdex

SUMMARY:
The goal of this proposal is to develop a more effective and better tolerated regimen. Ixazomib appears to have greater activity than bortezomib with less peripheral neuropathy.

DETAILED DESCRIPTION:
1.1 PRIMARY OBJECTIVE: 1.1.1 To evaluate the response rate of Ixazomib with metronomic cyclophosphamide and dexamethasone for first-line treatment of multiple myeloma 1.2 SECONDARY OBJECTIVES: 1.2.1To evaluate the toxicities associated with Ixazomib with metronomic cyclophosphamide and dexamethasone.

1.2.2 Estimate the progression-free survival and overall survival of Ixazomib with metronomic cyclophosphamide and dexamethasone for first-line treatment of multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Histologically confirmed multiple myeloma according to WHO classification. Pathology report to be sent to BrUOG for confirmation
* Diagnosis of Multiple Myeloma that has not been previously treated (although patients that received emergent steroid and/or local radiation therapy will be permitted to enter the study). , Details need to be submitted to BrUOG with dates and doses.
* Measureable disease defined as either an elevated serum M-protein, urine M-protein, bone marrow involvement >30% or serum free light chains per the IMWG criteria. Confirmation to be sent to BrUOG, see section 7 for criteria
* Life expectancy of ≥ 6 months, confirmation per treating investigator required
* Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment. If transfusional support provided, please document for submission to BrUOG
* Calculated creatinine clearance ≥30 mL/min (based on the Cockcroft-Gault Equation below)

For males:

Creatinine Clearance = (140-age[years] x weight [kg]) 72 x (serum creatinine[mg/dL])

For females:

Creatinine Clearance = 0.85 (140-age[years] x weight [kg]) 72 x (serum creatinine[mg/dL])

* ECOG performance status of 0-1.
* Adequate Liver function; AST or ALT < 3.0 x upper limit of normal (ULN); Total bilirubin <1.5x ULN
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug and obtain a pregnancy test, which must come back negative prior to drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject and obtain a serum pregnancy test, which must come back negative prior to drug. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.) Documentation and confirmation of conversations and patient commitment to contraception is required to be noted and sent to BrUOG. Female's menopausal status to be documented and submitted to BrUOG if applicable. Pregnancy test, if applicable, required to be sent to BrUOG.
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.) Documentation and confirmation of conversations and patient commitment to contraception is required to be noted and sent to BrUOG.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Any surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment.
* Central nervous system involvement (myeloma-related).
* Active infection requiring systemic antibiotic therapy or other serious active infection within 7 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol. If not applicable, then investigator to document not applicable
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent. If not applicable, then investigator to document not applicable
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing. If not applicable, then investigator to document not applicable
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has ≥ Grade 2 peripheral neuropathy or Grade 1 with pain.
* Participation in other therapeutic clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2019-03-29 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG
Locations (3):
- United States (3):
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Pelcovits A, Barth P, Reagan JL, Olszewski AJ, Rosati V, Wood R, Sturtevant A, Winer ES. Ixazomib, Oral Metronomic Cyclophosphamide, and Dexamethasone for First-Line Treatment of Multiple Myeloma: A Phase II Brown University Oncology Group Study. Oncologist. 2023 May 8;28(5):462-e303. doi: 10.1093/oncolo/oyad017. PMID 36942937

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixazomib Regimen: Cycle 1: Ixazomib: 4mg/day 1, 8, 15, Cyclophosphamide: 50 mg/day continuous daily, Dexamethasone: 20 mg/day 1, 8, 15 Cycles 2-6: Ixazomib: 4mg/day 1, 4, 8, 11, 15, 18, Cyclophosphamide: 50 mg/day continuous, daily, Dexamethasone: 20 mg/day 1, 4, 8, 11, 15, 18
  Maintenance:
  Ixazomib at 4 mg days 1, 8 and 15 of a 28 day cycle for 1 ½ years
  Ixazomib: Cycle 1:
  Ixazomib: 4mg/day 1, 8, 15
  Cycles 2-6:
  Ixazomib: 4mg/day 1, 4, 8, 11, 15, 18,
  Maintenance:
  Ixazomib at 4 mg days 1, 8 and 15 of a 28 day cycle for 1 ½ years
  Cyclophosphamide: Cycle 1:
  Cyclophosphamide: 50 mg/day continuous daily
  Cycles 2-6:
  Cyclophosphamide: 50 mg/day continuous daily
  Dexamethasone: Cycle 1:
  Dexamethasone: 20 mg/day 1, 8, 15
  Cycles 2-6:
  Dexamethasone: 20 mg/day 1, 4, 8, 11, 15, 18
Period: Overall Study
Arm/Group | Ixazomib Regimen
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib Regimen
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 61 [42 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Response Rate of Ixazomib With Metronomic Cyclophosphamide and Dexamethasone for First-line Treatment of Multiple Myeloma.
Time Frame: Through study treatment completion, an average of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Regimen
Number analyzed (Participants) | 12
Participants | 12

2. Secondary Outcome: Evaluation of the Toxicities Associated With Ixazomib With Metronomic Cyclophosphamide and Dexamethasone.
Time Frame: Assessed at baseline and end of study, up to 2 years, end of study reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Regimen
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: All adverse events and special reporting situations were reported from the time a signed and dated ICF is obtained until 30 days after the last dose of drug, up to 25 months, or until the subject withdraws consent from study participation (declines participation) or at the time patient becomes a screen failure, whichever occurs first, an average of 2 years.
Arm/Group | Ixazomib Regimen
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib Regimen (N=12)
Enterocolitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib Regimen (N=12)
Anemia (Blood and lymphatic system disorders) | 9
Palpitations (Cardiac disorders) | 1
Eye disorders, other (Eye disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Oral pain (Gastrointestinal disorders) | 1
Vomit (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Edema (General disorders) | 4
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Flu-like symptoms (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 7
Allergic reaction (Immune system disorders) | 1
Infection and infestations, other (Infections and infestations) | 6 — Flu
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 1
Creatinine increased (Investigations) | 6
Ejection fraction decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 11
Weight gain (Investigations) | 6
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasm benign, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Benign renal cyst
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7
Presyncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 6
Bladder pressure (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 10
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02412228/Prot_SAP_ICF_000.pdf